CLINICAL TRIAL: NCT02548741
Title: Evaluation of the Metformin Scavenging Mechanism on Methylglyoxal in Patients With Type 2 Diabetes Mellitus
Brief Title: Evaluation of the Metformin Effect on Methylglyoxal in Patients With Type 2 Diabetes
Acronym: MET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Serrine S. Lau, Professor, Department of Pharmacology and Toxicology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1506912530
Record Dates: First submitted 2015-08-24; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Metformin; diabetes; type 2 diabetes; diabetes complications; methylglyoxal; Prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetes Complications; Prediabetic State | interventions — Metformin; Calcium Carbonate; Urine Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Treatment (Metformin) (Active Comparator): Forty patients with elevated glycosylated hemoglobin A1c (HbA1c) > 6.0% (patients with type 2 diabetes mellitus or prediabetes) but HbA1C < 9.0%. They will receive the active comparator (metformin).
  Interventions: Drug: Metformin Hydrochloride (500-mg capsule); Other: Glucometer (One Touch glucometer), strips and lancets; Other: Urine container for 24-hour urine collection
- Placebo (Placebo Comparator): Forty patients with elevated glycosylated hemoglobin A1c (HbA1c) > 6.0% (patients with type 2 diabetes mellitus or prediabetes) but HbA1C < 9.0%. They will receive the placebo comparator.
  Interventions: Drug: Calcium carbonate (placebo); Other: Glucometer (One Touch glucometer), strips and lancets; Other: Urine container for 24-hour urine collection
- Non-diabetic (Other): Forty matched non-diabetic patients with HbA1C ≤ 5.6%. They will not receive either treatment (metformin) or placebo.
  Interventions: Other: Urine container for 24-hour urine collection

INTERVENTIONS:
Drug: Metformin Hydrochloride (500-mg capsule) — Metformin hydrochloride tablets (500-mg) are manufactured by Heritage Pharma INC. Noha Ashy & David Lee will ground the tablets and put them in capsules to avoid differentiation between treatment and placebo. Using USP 797 compounding standers, Noha Ashy & David Lee will package the capsules to conceal it from the participants and other investigators. Compounding will take place at the lab, College of Pharmacy (Darchman building, 2nd floor), University of Arizona. New empty capsules (size 0, ½ blue-opaque and ½ white-opaque capsule which will be supplied by Letco Medical) will be provided to the treatment (metformin hydrochloride) arm participants that are similar to the placebo (comparator) capsules in term of color and size to conceal placebo from the investigators and participants.
  Arms: Treatment (Metformin)
Drug: Calcium carbonate (placebo) — Investigators will use powder of calcium carbonate as filler of placebo capsules. Placebo capsules (size 0,½ blue-opaque and ½white-opaque capsule which will be supplied by Letco Medical),will be provided to the comparator arms' participants that are similar to the metformin hydrochloride capsules in term of color and size to conceal placebo from the investigators and participants.Using USP 797 compounding standers, Noha Ashy & David Lee will package the capsules to conceal it from the participants and other investigators. Compounding will take place at the lab, College of Pharmacy (Darchman building, 2nd floor), University of Arizona.
  Arms: Placebo
Other: Glucometer (One Touch glucometer), strips and lancets — Investigators will provide glucometer (One Touch glucometer), strips and lancets to the treatment and placebo groups. They will be provided to patients who never had glucometer before enrolling to our study.Also, a logbook will be provided to each participant to record their blood sugar measurements at home.
  Arms: Placebo; Treatment (Metformin)
Other: Urine container for 24-hour urine collection — During visit 2 (day 0) and visit 3 (day 42), urine container will be provided to the study participant for 24-hour urine collection. Patient will be instructed to bring the container back to the collaboratory. Investigators will transfer the urine container to Dr.Lau's lab to measure the IMZ concentration/content.

SUMMARY:
This study is designed to investigate the effects of metformin, a commonly prescribed first line medication for diabetes and recommended for prediabetes, on the levels of the potentially tissue damaging reactive product (MG) in the blood and its cleared counterpart in the urine (IMZ). The study will involve patients with elevated HbA1c randomized to receive either metformin or a similar inactive placebo pill and a group of sex and age matched volunteers without diabetes. Study participants will be recruited from the University of Arizona Medical Center, South Campus clinics (Endocrine clinic, family medicine clinic and general medicine clinic). Eighty patients with HbA1c >6.0% will be randomized to receive either metformin or a similar inactive placebo for 6 weeks. The response of these patients will be compared to 40 patients normal HbA1c <5.6% who will not receive either study medication. Investigators will compare the plasma MG and urine IMZ concentration/content between the 3 groups before and after the 6-week intervention. It is hypothesized that plasma MG level in the metformin treatment group will be less than in the group taking the placebo pills, while there will be no significant difference in MG level between the metformin treatment group and the volunteers without diabetes.

DETAILED DESCRIPTION:
A prospective randomized controlled clinical trial of 120 adult patients will be conducted from June 2015 to June 2017 (2 years). Study participants will be recruited from the University of Arizona Medical Center, South Campus clinics (Endocrine clinic, family medicine clinic and general medicine clinic).

Eighty patients with HbA1c* >6.0% will be randomized to receive either metformin or a similar inactive placebo for 6 weeks. The response of these patients will be compared to 40 patients with normal HbA1c <5.6% who will not receive either study medication.

Twenty four-hour urine samples will be analyzed to measure metformin-MG adducted product (IMZ) at baseline (D0) and at the end of the study period (D42). Blood sample will be analyzed at the baseline to measure the plasma methylglyoxal concentration (baseline MG concentration- D0) and re-measure it at the end of the study period(D42). Mass spectrometry will be performed for samples analysis to detect the plasma methylglyoxal (MG) level. Metformin-MG adducted product (IMZ) will be measured using Multiple Reaction Method (MRM). Also, Mass spectrometry will be performed to detect plasma protein modifications at baseline and at the end of the study period (after 6 weeks). Investigators will measure the concentrations of IMZ and MG in the human urine and plasma of our cohort in the nM and μM range, respectively via mass spectrometry. Investigators will be normalizing these values by specific gravity.

A logbook will be provided to each participant to record their blood sugar measurements at home. Investigators will provide glucometer (One Touch glucometer), strips and lancets to patients who never had glucometer before enrolling to our study. Participants taking metformin or placebo will be asked to perform an 4-point self-measured blood sugar profile with measurements taken as indicated in the table (once a week). Investigators will contact study participants (treatment and placebo group only) by phone at the mid of the study period (D21) to follow up on the recorded fasting blood glucose levels and development of side effects. The results of the blood sugar measurements will help the study physicians to adjust diabetes therapy (metformin or the other concomitant diabetes medications) in order that the study subjects maintain appropriate blood glucose control (target pre-meal and bedtime glucose between 90-180 mg/dL).

The participants in the non-diabetic group, they will not receive either metformin hydrochloride or placebo. Their fasting blood glucose, plasma MG level and urine IMZ level will be measured during the study. They will not be required to perform 4 point testing. They will have all the same clinic visits and lab orders as diabetic patients except receiving the study medication.

It is hypothesized that plasma MG level in the metformin treatment group will be less than in the group taking the placebo pills, while there will be no significant difference in MG level between the metformin treatment group and the volunteers without diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Elevated HbA1c > 6.0% (patients with type 2 diabetes mellitus or prediabetes), HbA1C < 9.0%
* For matched non-diabetic patients: HbA1C ≤ 5.6%
* Serum creatinine (SCr) < 1.5 mg/dL in males or < 1.4 mg/dL in females,
* Calculated glomerular filtration rate (GFR) > 60 ml/min/1.73m2,
* Body mass index (BMI) 25-40 kg/m2,
* Glycosylated hemoglobin A1C (HA1C) < 9%,
* No known intolerance to metformin
* Has not taken metformin previous 3 months

Exclusion Criteria:

* Patients on thiazolidinediones (TZD)
* Patients with history of metformin intolerance (gastrointestinal side effects or poor renal function; Serum Cr > 1.5mg/dL in males or > 1.4 mg/dL in females or calculated GFR < 60 mL/min/1.73m2
* Patients with active (symptomatic or unstable) cardiovascular disease
* Patients requiring home oxygen
* Patients with end-stage liver disease (cirrhosis)
* Patients on oral glucocorticoids within the past 30 days (equivalent to prednisone > 5mg/day)
* Excessive alcohol intake (The Substance Abuse and Mental Health Services Administration (SAMHSA) defines heavy drinking as drinking 5 or more drinks on the same occasion on each of 5 or more days in the past 30 days) 29
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Plasma methylglyoxal (MG) concentration (μM) | Change from baseline in plasma MG concentration at 6 weeks of metformin administration
  Investigators will measure MG concentration at baseline and after 6 weeks of metformin administration. An increase in MG has been associated with type-2 diabetes and progression of diabetes complications. Metformin is a known scavenger of MG, forming a metformin-MG imidazolinone (IMZ) cyclized product. This unique property of metformin in enhanced reduction of diabetic complications may be related to its MG-scavenging capabilities. Investigators will measure the concentrations of MG in the human plasma of the cohort in the μM range via mass spectrometry. Investigators will be normalizing these values by specific gravity.

SECONDARY OUTCOMES:
The urine imidazolinone (IMZ) concentration (nM) | Change from baseline in urine IMZ concentration at 6 weeks of metformin administration
  Metformin is a known scavenger of MG, forming a metformin-MG imidazolinone (IMZ) cyclized product. This unique property of metformin in enhanced reduction of diabetic complications may be related to its MG-scavenging capabilities. Investigators will measure the IMZ concentration/content at baseline and after 6 weeks of metformin administration. Investigators hypothesized that a concomitant elevation in urine IMZ concentration/content is associated with metformin administration. Investigators will measure the concentrations of IMZ in the human urine plasma of the cohort in the nM range via mass spectrometry. Investigators will be normalizing these values by specific gravity.

CONTACTS AND LOCATIONS:
Overall Officials: Serrine S Lau, PhD, Principal Investigator — University of Arizona; Craig Stump, MD, PhD, Study Director — University of Arizona